CLINICAL TRIAL: NCT04767321
Title: A Phase I/IIa, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety and Exploratory Efficacy of 3% LTX-109 Compared to Placebo for Nasal Decolonisation of Staphylococcus Aureus
Brief Title: A Study to Evaluate the Safety and Efficacy of 3% LTX-109 for Nasal Decolonisation of Staphylococcus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pharma Holdings AS (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C20-109-06
Record Dates: First submitted 2021-02-12; First posted 2021-02-23 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-02

CONDITIONS: Nasal Decolonization of Staphylococcus Aureus

STUDY DESIGN:
Intervention Model Description: Randomised, Double-blind, Placebo-controlled Randomization 3:1, active to placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTX-109 treatment (Experimental): Nasal application of LTX-109 gel 3% (w/w), 250 mikroliters in each nostril, 4 times in one day, every two hours.
  Interventions: Drug: LTX-109 gel, 3% w/w
- Placebo (Experimental): Nasal application of placebo, 250 mikroliters in each nostril, 4 times in one day, every two hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LTX-109 gel, 3% w/w — LTX-109 gel will be applied topically to both nostrils by a qualified health professional. On each dosing occasion, a large drop of IMP will be applied into each nostril and distributed to cover the whole area of the nostril.
  Arms: LTX-109 treatment
Drug: Placebo — Placebo gel will be applied topically to both nostrils by a qualified health professional. On each dosing occasion, a large drop of IMP will be applied into each nostril and distributed to cover the whole area of the nostril.
  Arms: Placebo

SUMMARY:
A Phase I/IIa, double-blind, placebo-controlled, randomised study designed to evaluate the safety, tolerability, exploratory efficacy and exposure of LTX-109 administered topically to the anterior nares in subjects with persistent carriage of S. aureus (methicillin-susceptible S. aureus [MSSA] and/or methicillin-resistant S. aureus [MRSA]).

DETAILED DESCRIPTION:
Approximately 60 subjects will be screened to achieve 24 persistent MSSA and/or MRSA carriers and 16 randomised and dosed subjects randomized 3:1, active to placebo.

Eligible subjects will be admitted to the clinic on Day 1 for randomisation and dosing and will remain at the clinic until Day 2. Following nasal and perineum swabs and a chlorhexidine (Hibiscrub®) shower, the investigational medicinal product (IMP) will be applied topically to both nostrils by a qualified health professional 4 times during a six hour period (every two hours at 0, 2, 4 and 6 hours) on Day 1.

Subjects will come back to the research clinic on Day 3, Day 4, Day 8 and Day 15 (Visits 4 to 7) for safety, tolerability and efficacy assessments and for blood sampling for bioanalysis. On Day 5 and Day 6, subjects will take a chlorhexidine shower at home. A final end-of-study visit (Visit 8) will take place on Day 22 (±3 days) or after early withdrawal.

All subjects will be instructed to wash the body and hair with chlorhexidine body wash and shampoo at the clinic on Day 1 (prior to the first dose) and on Day 2. Prior to leaving the clinic on Day 2, subjects will be provided with chlorhexidine body wash and shampoo for body and hair wash at home on Day 3 (prior to Visit 4), on Day 4 (prior to Visit 5) and on Day 5 and Day 6.

Each subject is expected to participate in the study for approximately 50 days including a 28 day screening period

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Male or female subject aged 18 to 65 years inclusive at Visit 2.
3. Persistent nasal carrier of Staphylococcus aureus (MSSA and/or MRSA), confirmed by two positive bacterial cultures from the nose during the screening period.
4. Clinically normal medical history, physical findings, vital signs and laboratory values at the time of screening Visit 2, as judged by the Investigator.
5. Women of child bearing potential (WOCBP) must practice abstinence (only allowed when this is the preferred and usual lifestyle of the subject) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]) from at least 2 weeks prior to dose to 2 weeks after last dose. Female subjects must refrain from donating eggs from the date of dosing until 3 months after dosing with the IMP. Their male partner must agree to use a condom during the same time frame if he has not undergone vasectomy.

Women of non-childbearing potential are defined as pre-menopausal females who are sterilised (tubal ligation or permanent bilateral occlusion of fallopian tubes); or females who have undergone hysterectomy or bilateral oophorectomy; or post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with simultaneous detection of follicle stimulating hormone [FSH] 25-140 IE/L is confirmatory).

Male subjects must be willing to use condom or be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the date of dosing until 3 months after dosing with the IMP. Their female partner of child-bearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above).

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
3. Severe eczema or skin wounds, dry or sensitive skin assessed as clinically significant by the Investigator.
4. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
5. Any positive result at screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
6. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to LTX-109 or chlorhexidine.
7. S. aureus (MSSA and/or MRSA) decolonisation attempt in the 6 months prior to screening Visit 2.
8. Inability to take medications nasally.
9. Nasal polyps or significant anatomical nasal abnormality, as judged by the Investigator.
10. Evidence of open wound, lesion, inflammation, erythema or infection (including active rhinitis, sinusitis or upper respiratory infection) affecting the nostril area, lip and skin close to the nose.
11. History of multiple episodes (>3) of epistaxis within 12 months prior to screening Visit 2.
12. Disease in the region of the application sites, significant history of trauma or skin disease in the region of the application sites, current nasal skin or nasal septum condition requiring treatment or nasal surgery in the 6 months prior to screening Visit 2.
13. In situ nasal jewellery or open nasal piercings.
14. Previous or concurrent treatment with antimicrobials for an infection within the last 30 days prior to the first administration of IMP.
15. Regular use of cortisone or anticoagulation medication within 14 days prior to the first administration of IMP and regular use of nasal decongestants within 30 days prior to the first IMP administration, at the discretion of the Investigator.
16. Planned treatment or treatment with another investigational drug within 30 days prior to Day 1. Subjects consented and screened but not dosed in previous Phase I studies are not excluded.
17. Positive screen for drugs of abuse or alcohol at screening Visit 2 or on admission to the unit prior to administration of the IMP.
18. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
19. Presence or history of drug abuse, as judged by the Investigator.
20. History of, or current use of, anabolic steroids.
21. Plasma donation within 2 weeks of screening Visit 2 or blood donation (or corresponding blood loss) during the three months prior to screening.
22. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.
23. Female subjects who are pregnant or who are currently breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of safety by occurence and frequency of Adverse Events | Through treatment and followup of 22 days
  Occurrence and frequency of Adverse Events
Local tolerability assessed by a qualified health care professional by evaluation of nostrils and scoring using a 4-point graded scale. | Day 1
  Incidence of local reactions (erythema, swelling and lesions) will be assessed by a qualified health care professional . Each nostril will be evaluated separately and scored using a 4-graded scale (0-3)
Local tolerability assessed by a qualified health care professional by evaluation of nostrils and scoring using a 4-point graded scale. | Day 2
  Incidence of local reactions (erythema, swelling and lesions) will be assessed by a qualified health care professional . Each nostril will be evaluated separately and scored using a 4-graded scale (0-3)
Local tolerability assessed by a qualified health care professional by evaluation of nostrils and scoring using a 4-point scale. | Day 3
  Incidence of local reactions (erythema, swelling and lesions) will be assessed by a qualified health care professional . Each nostril will be evaluated separately and scored using a 4-graded scale (0-3)
Local tolerability assessed by a qualified health care professional by evaluation of nostrils and scoring using a 4-point scale. | Day 4
  Incidence of local reactions (erythema, swelling and lesions) will be assessed by a qualified health care professional . Each nostril will be evaluated separately and scored using a 4-graded scale (0-3)
Local tolerability assessed by a qualified health care professional by evaluation of nostrils and scoring using a 4-point scale. | Day 8
  Incidence of local reactions (erythema, swelling and lesions) will be assessed by a qualified health care professional . Each nostril will be evaluated separately and scored using a 4-graded scale (0-3)
Local tolerability assessed by a qualified health care professional by evaluation of nostrils and scoring using a 4-point scale. | Day 15
  Incidence of local reactions (erythema, swelling and lesions) will be assessed by a qualified health care professional . Each nostril will be evaluated separately and scored using a 4-graded scale (0-3)
Local tolerability assessed by a qualified health care professional by evaluation of nostrils and scoring using a 4-point scale. | Day 22
  Incidence of local reactions (erythema, swelling and lesions) will be assessed by a qualified health care professional . Each nostril will be evaluated separately and scored using a 4-graded scale (0-3)
Local tolerability assessed by the subject by Visual Analog Scale. | Day 1
  Assessment of Local tolerability on Visual Analog Scale
Local tolerability assessed by the subject by Visual Analog Scale. | Day 2
  Assessment of Local tolerability on Visual Analog Scale

SECONDARY OUTCOMES:
Number of subjects on LTX-109 versus placebo with bacterial eradication at Test of Cure | 54 hours (+ 2 hours)
  Assessment of eradication of bacteria defined as non-presence of Staphylococcus aureus (MSSA and/or MRSA) in quantitative cultures
Number of subjects on LTX-109 versus placebo with bacterial eradication at other specified time points than Time of Cure. | 4, 6, 12, 24, 78 hours and Days 8, 15 and 22
  Assessment of bacterial count at specified points in time to explore effect of the intervention
Number of colony forming units (CFUs) in subjects on LTX-109 versus placebo at specified points in time. | 4, 6, 12, 24, 78 hours and Days 8, 15 and 22
  Assessment of bacterial count at specified points in time to explore effect of the intervention
Number of subjects on LTX-109 vs placebo with bacterial recolonisation defined as the timepoint of recurrence of colonisation after confirmed eradication. | Days 4, 8, 15 and 22
  Assessment of recurrence
Plasma concentrations of LTX-109 | 6, 24, 54 and 78 hours
  Assessment of plasma concentratin by analysis of blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Johan Nilsson, MD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- ClinSmart Sweden AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No